CLINICAL TRIAL: NCT05207917
Title: How Gastric Bypass and Sleeve Gastrectomy Change Social Experiences and Biomarkers of Well-being
Brief Title: How Does Bariatric Surgery Affect Social Experiences and Well-being - The BaSES-study
Acronym: BaSES
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Professor, The Hospital of Vestfold
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 238406
Record Dates: First submitted 2021-12-08; First posted 2022-01-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: 2 intervention groups with either sleeve gastrectomy (SG) or Roux-en-Y gastric bypass (RYGB) surgery; in addition one small exploratory group undergoing undergoing single anastomosis sleeve ileal (SASI) bypass
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastric bypass (Active Comparator): Gastric bypass
  Interventions: Procedure: Gastric bypass
- Sleeve gastrectomy (Active Comparator): Sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- Single anastomosis sleeve ileal (SASI) bypass (Experimental): Exploratory small arm with a small number of particpants
  Interventions: Procedure: Single anastomosis sleeve ileal (SASI) bypass

INTERVENTIONS:
Procedure: Gastric bypass — In Roux-en-Y gastric bypass (RYGB), the left crus will be dissected free, any hiatal hernia left in place. The minor curvature is opened at the second vessel and the lesser sac entered. A 25 mL gastric pouch will be created by firing one horizontal and two vertical staple loads. The ligament of Treitz is then identified and a proximal loop of small intestine anastomosed to the pouch 60 cm from the ligament of Treitz with one linear stapler (full length of the stapler), creating an antecolic, antegastric alimentary limb. The opening will be closed using a single row, running absorbable suture. An entero-enteroanastomosis will be made 120 cm distal of the gastro-enteroanastomosis. The introductory opening is closed with a single row, running absorbable suture. The small intestine will be divided with one load between the gastro-entero-enteroanastomosis and the entero-enteroanastomosis in order to complete a bypass with an alimentary limb of 120 cm and a biliopancreatic limb of 60 cm.
  Arms: Gastric bypass
Procedure: Sleeve gastrectomy — In sleeve gastrectomy (SG) a large part (80%) of the ventricle is removed. The greater curvature will be dissected free starting 4-5 cm from the pylorus up to the angle of Hiss. The left crus is then visualized and inspected for hiatal hernia. Small sliding hernias and wide hiatus are left in situ. The ventricle will then be lifted and any adhesions in the lesser sac divided. A 35 Fr bougie is placed down to the pylorus guiding the creation of a tubular sleeve with linear staplers. The first two loads are always green or purple, while blue or tan loads are used for the rest of the ventricle. The last stapler is placed 5 mm laterally to the angle of Hiss. The staple line will then be inspected and secured with clips for additional haemostasis, no oversewing or buttressing material is routinely used.
  Arms: Sleeve gastrectomy
Procedure: Single anastomosis sleeve ileal (SASI) bypass — The SASI bypass will performed with a similar entry of the abdominal cavity. A 6-port set up and a liver retractor is utilized. The small bowel is measured 300cm from the ileocecal valve, in sequences of 10cm, with the small bowel stretched and markers placed on the graspers, and connected to the antrum of the stomach with a 45mm stapler. The anastomosis is positioned slightly ventral on the antrum. The antrum is opened ventrally 5 cm proximal to the pylorus, just below the horizontal axis of canalis pylori. A 12 mm port positioned left to the midline is used for introduction of the stapler, which is directed distally from the patient's left to right side. 2.5 cm of the 45 mm stapler device is used for firing the anastomosis, which is completed with a 2-0 PDS running suture. The fascia defect is closed for the port where the specimen is extracted. The mesenteric defect is not closed.
  Arms: Single anastomosis sleeve ileal (SASI) bypass

SUMMARY:
Nonrandomized controlled trial to assess whether or not sleeve gastrectomy (SG) or Roux-en-Y gastric bypass (RYGB) affect social experiences and biomarkers of well-being 6 weeks and 1 year after surgery. The decision whether SG or RYGB will be performed is determined by medical decision making. Hypotheses: Bariatric surgery influences social experiences and well-being through changes in body image, reward responsivity and gut hormones. These changes may differ between gastric bypass (RYGB) and sleeve gastrectomy (SG).

DETAILED DESCRIPTION:
Explanation for choice of comparators

Obesity is one of the world's most serious public health problems. Conservative weight reduction methods alone (diet, exercise) often show disappointing results, as the majority of people who lose weight regain it after a shorter or longer period of time. The currently most effective measure to achieve a durable weight-loss is bariatric surgery.

When investigating the effectiveness of bariatric surgery, the focus has most often been on weight loss and obesity-related complications, while effects on social interaction and subjective experience have received much less attention. A large body of evidence has demonstrated that (supportive) social relationships benefit health. Individuals with low compared to those with high levels of social connectedness are more likely to die prematurely; and social relationships can also affect a range of other health conditions such as cardiovascular disease, cancer, and immune function. Importantly, individuals with obesity may experience social interactions as less positive than normal-weight individuals. They recount avoiding social events and relationships, but also career opportunities, shopping and other activities where they feel observed because of weight stigma. Such avoidance behavior can lead to a "chronic disengagement" with many aspects of social life, which in turn might decrease interpersonal skills. Further investigations into the link between social behavior and eating found that greater emotional eating is associated with greater social avoidance. Eating was described a means to cope with loneliness on the one hand, while on the other hand aggravating feelings of being alone due to the stigma associated with obesity. This way, loneliness and obesity can create a vicious circle. In terms of how bariatric surgery influences social interactions, one 10-year follow up study found improvements in social interactions for bariatric surgery, but not for conventional weight loss treatment. In qualitative studies, many participants mentioned that they received more positive social feedback following bariatric surgery, and that they enjoyed social activities more than before, although they also describe ambiguous feelings.

The present study will investigate whether and how two types of bariatric surgery improve the response to a range of social aspects of patients' daily lives. Further, it aims to determine potential mechanisms leading to these effects, namely changes in body image, gut hormones, and reward responsivity.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for bariatric surgery and eligible for sleeve gastrectomy or gastric bypass
* able to give consent
* understand written and spoken Norwegian

Exclusion Criteria:

* pregnancy and breast-feeding
* chronic disease (endocrine, heart, neurological, lung, gastrointestinal, kidney)
* cancer
* acute psychotic episode

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
1-year changes in Social Experience | Change from 4 weeks before surgery to 1 year after surgery
  10-item checklist assessing frequency and quality of daily social interactions (preprint in August 2025: https://osf.io/preprints/psyarxiv/6psar_v2); 2 sub-scales: (1) Being with others, (2) Being alone; the diary will be filled in 14 days in a row at the end of the day. Scale (1) was designed to measure enjoyment of being with others and the duration of social contact (6 items, range: 4 to 62.4), higher values indicate more enjoyment and a higher frequency of social contact. Scale (2) was designed to measure enjoyment of being alone (3 items, range: -5 to 20), higher values here indicate more enjoyment of being alone. An additional item at the beginning of the checklists asks how many people the respondent has had social contact with during the day (5 categories).

SECONDARY OUTCOMES:
Changes in affect ratings after social evaluation (inclusion and exclusion) | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Positive and Negative Affect Schedule (PANAS): The PANAS is a self-report measure that is made up of two mood scales of 10 adjectives each, one measuring positive affect and the other one measuring negative affect. (1) Positive Affect Scale (range: 10-50; higher values indicate higher positive affect); (2) Negative Affect Scale (range: 10-50, higher values indicate higher negative affect)
Changes in experience ratings after social evaluation (inclusion and exclusion) | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Need-Threat Scale: 4 sub-scales: (1) Belonging, (2) Self-Esteem, (3) Meaningful existence, (4) Control; range: 3-27 per sub-scale; higher values indicate more belonging, higher self-esteem, higher meaningful existence, and more control)
Changes in pleasantness ratings in response to touch stimulation on the forearm | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Subjective ratings on a digitally presented visual analogue scale (VAS) scale: range 0-100 (unpleasant - pleasant) after a touch stimulation to the forearm (repeated 10 times)
Changes in pleasantness ratings in response to self-stroking on the forearm | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Subjective ratings on a digitally presented VAS scale: range 0-100 (unpleasant - pleasant), after participants made 10 back-and-forth strokes on their forearm with their hand
Changes in intensity ratings in response to touch stimulation on the forearm | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Subjective ratings on a digitally presented VAS scale: range 0-100 (not intense - intense), after a touch stimulation to the forearm (repeated 10 times)
Changes in intensity ratings in response to self-stroking on the forearm | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Subjective ratings on a digitally presented VAS scale: range 0-100 (not intense - intense), after participants made 10 back-and-forth strokes on their forearm with their hand
Changes in self-stroking velocity | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Participants are instructed to stroke their own forearm with a velocity they experience as pleasant. The duration of 10 back-and-forth strokes over a 10 cm distance on the forearm will be measured with a stop watch. Velocity in cm/sec will be calculated thereafter.
Changes in cortisol levels from hair samples | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Cortisol (in pg/mg)
Changes in endocannabinoid levels from hair samples | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Endocannabinoids (in pg/mg)
Changes in fasting ghrelin levels from blood samples | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Ghrelin (in pg/ml)
Changes in body image | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaires: Appearance Evaluation Scale (AES) and the Body Areas Satisfaction Scale (BASS) - the AES was designed to measure overall satisfaction/dissatisfaction with one's appearance and physical attractiveness. It has 7 items (range: 5-35) with high scores indicating body satisfaction and low scores indicating body dissatisfaction. The BASS was designed to measure the degree of dissatisfaction-satisfaction with specific body areas and attributes (range: 9-45). Higher scores indicate greater body satisfaction and lower scores indicate greater body dissatisfaction.
Changes in reward responsivity | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire: Temporal Experience of Pleasure Scale (TEPS) - the TEPS was designed to measure individual trait dispositions in both anticipatory and consummatory experiences of pleasure. It consists of 18 items, of which 10 form the (1) anticipatory pleasure scale (range: 10-60), and (2) 8 items for the consummatory pleasure scale (range: 8-48). Higher values on (1) indicate enhanced reward responsiveness and imagery, while higher values on (2) indicate higher openness to different experiences and appreciation of positive stimuli.
Changes in interoceptive ability | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire: Body Awareness Questionnaire (BAQ) - the BAQ was designed to assess self-reported attentiveness to normal nonemotive body processes, such as sensitivity to body rhythms, ability to detect small changes in normal bodily functioning, and one's ability to anticipate bodily reactions. It consists of 18 items (range: 18-126). Higher values indicate a higher sensitivity and awareness of one's bodily states.
Changes in belongingness | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaires: The Social Connectedness Scale Revised (SCS-R) and the Social Assurance Scale (SAS). The SCS-R was designed to measure a psychological sense of belonging, or how individuals cognitively construe interpersonal closeness with others in their social world. It consists of 20 items (range: 20-120), with higher values indicating a higher sense of belonging. The SAS was designed to measure the importance of assurance from one's social group.It consists of 8 items (range: 8-48), with higher values indicating a higher need for social assurance.
Changes in social network size | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire: The Social Network Index (SNI) - the SNI was designed to measure three aspects of one's social networks: (1) network diversity, (2) number of people in the network, and (3) number of embedded networks. Each of the three sub-scales is assessed on 12 items. (1) refers to the number of high-contact roles (range: 0-12), with higher values indicating a higher number of social roles. (2) refers to the total number of people with whom the respondent has regular contact, which will be summed for the 12 items (range: 0-70). Higher numbers indicate more people in one's network (to not inflate the number, items 4-12 will be scored with 7 in case the reported number of people in this group is equivalent or larger to 7). The embedded network scale (3) reflects the number of different network domains in which a respondent is active (range: 0-8), with higher numbers indicating activity in more network domains.
Changes in self-reported eating patterns | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire:The Three Factor Eating Questionnaire -R 21 (TFEQ-R21) measures eating behaviour and has been validated for use in individuals with obesity and will be used in the study. It consists of 21 items comprising three domain scores; (1) uncontrolled eating; assessing the tendency to lose control over eating when feeling hungry or when exposed to external stimuli, (2) cognitive restraint; assessing the conscious restriction of food intake to control body weight or body shape, and (3) emotional eating; assessing overeating related to negative mood states. The domain scores were transformed to 0-100 scales to facilitate comparison; a higher score indicates more uncontrolled, restraint, or emotional eating.
Changes in symptoms of depression and anxiety | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire: Hospital Anxiety and Depression Scale (HADS). The validated generic HADS measures symptoms of anxiety and depression using 14 items scored from 0-3 It is decomposed into two domains measuring depression (HADS-D) and anxiety (HADS-A), both consisting of seven items yielding a score from 0-21.
Changes in Health Related Quality of Life 1 | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Generic questionnaire: Short Form-36 Health Survey (SF-36). Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores for each of the 8 domains and summary scores for physical and mental health will be calculated.
Changes in Health Related Quality of Life 2 | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Questionnaire: Weight-related Symptom Measure (WRSM). The validated obesity specific WRSM measures 20 symptoms commonly related to being overweight or obese, including foot problems, joint pain, sensitivity to cold, shortness of breath, etc. using two different sets of items. The first set assesses whether or not a patient is experiencing specific symptoms, and the second set rates the level of the distress of the symptoms with values from zero ("not at all") to six ("bothers a very great deal"). The first set creates an additive scale summing symptoms from 0-20, while the second forms a symptom distress scale ranging from 0-120.
Changes in Health Related Quality of Life 3 | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Obesity specific questionnaire: The Impact of Weight on Quality of Life-Lite (IWQOL-lite). The IWQOL-Lite is a 31-item measure of weight-related quality of life. There are five domain scores (Physical Function, Self-Esteem, Sexual Life, Public Distress and Work) and a total score. Scores for all domains and total score range from 0-100, with lower scores indicating greater impairment.
6-week Changes in Social Experience | Change from 4 weeks before surgery to 6 weeks after surgery
  10-item checklist assessing frequency and quality of daily social interactions (preprint in August 2025: https://osf.io/preprints/psyarxiv/6psar_v2); 2 sub-scales: (1) Being with others, (2) Being alone; the diary will be filled in 14 days in a row at the end of the day. Scale (1) was designed to measure enjoyment of being with others and the duration of social contact (6 items, range: 4 to 62.4), higher values indicate more enjoyment and a higher frequency of social contact. Scale (2) was designed to measure enjoyment of being alone (3 items, range: -5 to 20), higher values here indicate more enjoyment of being alone. An additional item at the beginning of the checklists asks how many people the respondent has had social contact with during the day (5 categories).
Group differences between SG and RYBG patients in the above-mentioned outcomes [1-22] | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  The above-mentioned outcomes will be tested for differences between the two surgery types.

OTHER OUTCOMES:
Change in Body Mass Index (BMI) | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  calculated from height (in cm) and weight (in kg) as kg/m^2
Change in weight | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Percent total weight loss (%TWL) and in kg
Change in anthropometric measures | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Waist and hip circumference (cm)
Change in body fat | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Body fat (in %)
Change in fat-free mass | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Fat-free mass (in kg)
Change in blood pressure | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Systolic and diastolic blood pressure (mm/Hg)
Change in lipids | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Total-cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides (all in mmol/l)
Change in glucose parameters | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  HbA1c (mmol/mol); C-peptide (nmol/l)
Change in C-reactive protein (CRP) | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  CRP (mg/L)
Change in blood enzymes | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  ASAT (aspartate aminotransferase), ALAT (alanine-aminotransferase), LD (lactate dehydrogenase), Gamma-GT (gamma-glutamyl transferase), ALP (alkaline phosphatase) (all in U/L)
Change in hemoglobin | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Hemoglobin (g/100 ml)
Change in ferritin | Change from 4 weeks before surgery to 6 weeks and 1 year after surgery
  Ferritin ((µg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, Professor, Principal Investigator — The Hospital of Vestfold
Locations (1):
- Morbid Obesity Center, Tønsberg, Vestfold, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-anonymized individual participant data can be made available following publication upon reasonable request to authors Jøran Hjelmesæth and Uta Sailer. Data will be shared according to the consent given by the participants and Norwegian laws and legislation.
Time Frame: For at least 10 years after publication
Access Criteria: All requests must be handled within the legal framework of Norway; non-commercial use of de-anonymized data

REFERENCES:
- [Background] Broadhead WE, Kaplan BH, James SA, Wagner EH, Schoenbach VJ, Grimson R, Heyden S, Tibblin G, Gehlbach SH. The epidemiologic evidence for a relationship between social support and health. Am J Epidemiol. 1983 May;117(5):521-37. doi: 10.1093/oxfordjournals.aje.a113575. No abstract available. PMID 6342368
- [Background] Uchino BN. Social support and health: a review of physiological processes potentially underlying links to disease outcomes. J Behav Med. 2006 Aug;29(4):377-87. doi: 10.1007/s10865-006-9056-5. Epub 2006 Jun 7. PMID 16758315
- [Background] Umberson D, Montez JK. Social relationships and health: a flashpoint for health policy. J Health Soc Behav. 2010;51 Suppl(Suppl):S54-66. doi: 10.1177/0022146510383501. PMID 20943583
- [Background] Maphis LE, Martz DM, Bergman SS, Curtin LA, Webb RM. Body size dissatisfaction and avoidance behavior: how gender, age, ethnicity, and relative clothing size predict what some won't try. Body Image. 2013 Jun;10(3):361-8. doi: 10.1016/j.bodyim.2013.02.003. Epub 2013 Mar 27. PMID 23540887
- [Background] Brytek-Matera A, Czepczor-Bernat K, Olejniczak D. Food-related behaviours among individuals with overweight/obesity and normal body weight. Nutr J. 2018 Oct 16;17(1):93. doi: 10.1186/s12937-018-0401-7. PMID 30326901
- [Background] Karlsson J, Taft C, Ryden A, Sjostrom L, Sullivan M. Ten-year trends in health-related quality of life after surgical and conventional treatment for severe obesity: the SOS intervention study. Int J Obes (Lond). 2007 Aug;31(8):1248-61. doi: 10.1038/sj.ijo.0803573. Epub 2007 Mar 13. PMID 17356530
- [Background] Coulman KD, MacKichan F, Blazeby JM, Owen-Smith A. Patient experiences of outcomes of bariatric surgery: a systematic review and qualitative synthesis. Obes Rev. 2017 May;18(5):547-559. doi: 10.1111/obr.12518. Epub 2017 Mar 8. PMID 28273694
- [Derived] Pfabigan DM, Hertel JK, Svanevik M, Lindberg M, Sailer U, Hjelmesaeth J. Single-centre, non-randomised clinical trial at a tertiary care centre to investigate 1-year changes in social experiences and biomarkers of well-being after bariatric surgery in individuals with severe obesity: protocol for the Bariatric Surgery and Social Experiences (BaSES) study. BMJ Open. 2023 Aug 28;13(8):e071332. doi: 10.1136/bmjopen-2022-071332. PMID 37640458